CLINICAL TRIAL: NCT03616392
Title: A Randomized, Open-label, Multiple Dose, 2-way Crossover Study to Evaluate the Drug Drug Interaction of CKD-501 and D308 in Healthy Volunteers
Brief Title: Clinical Trial to Evaluate the Drug Drug Interaction of CKD-501 and D308
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 19DDI18013
Record Dates: First submitted 2018-07-08; First posted 2018-08-06 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Diabetes Mellitus, Type II
Keywords: Diabetes Mellitus, Type II
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lobeglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part 1: Group 1(Treatment A/Treatment B) (Experimental): Period 1: Treatment A (D308 1T)/day for 5days, QD, PO Period 2: Treatment B (D308 1T + CKD-501 1T)/day for 5days, QD, PO
  Interventions: Drug: D308, CKD-501
- Part 1: Group 2(Treatment B/Treatment A) (Experimental): Period 1: Treatment B (D308 1T + CKD-501 1T)/day for 5days, QD, PO Period 2: Treatment A (D308 1T)/day for 5days, QD, PO
  Interventions: Drug: D308, CKD-501
- Part 2: Group 1(Treatment C/Treatment B) (Experimental): Period 1: Treatment C (CKD-501 1T)/day for 5days, QD, PO Period 2: Treatment B (D308 1T + CKD-501 1T)/day for 5days, QD, PO
  Interventions: Drug: D308, CKD-501
- Part 2: Group 2(Treatment B/Treatment C) (Experimental): Period 1: Treatment B (D308 1T + CKD-501 1T)/day for 5days, QD, PO Period 2: Treatment C (CKD-501 1T)/day for 5days, QD, PO
  Interventions: Drug: D308, CKD-501

INTERVENTIONS:
Drug: D308, CKD-501 — 1. D308
  2. CKD-501: Lobeglitazone sulfate 0.5mg

SUMMARY:
Phase 1 trial to evaluate the drug drug interaction of CKD-501 and D308

DETAILED DESCRIPTION:
A randomized, open-label, multiple dose, 2-way crossover study to evaluate the drug drug interaction of CKD-501 and D308 in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult older than 19 years at the time of screening
2. BMI 17.5~30.5kg/m2 and body weight more than 55kg
3. Subject who has no chronic disease within last 3 years and no symptoms or pathological findings
4. Suitable subject who is determined to be suitable at the time of screening such as laboratory tests(hematology, blood chemistry, urinalysis, virus/bacteriological test, etc.), sign of vitality, electrocardiogram
5. Subject who signed the written consent of the Chonbuk National University Hospital IRB to participate in this study with full understanding of the purpose and contents of the examination prior to the clinical trial
6. Subject who has will and ability to participate in clinical trials

Exclusion Criteria:

1. Subject who has a history of clinical significant blood, kidney, endocrine, respiratory, gastrointestinal, urinary, cardiovascular, liver, psychiatric, neurological or allergic diseases(except for asymptomatic seasonal allergies not treated at the time of administration) or evidence(except for simple dental history such as dental calculus, impacted tooth, wisdom tooth, etc.)
2. Subject with a history of gastrointestinal disorders(esophageal achalasia or esophagus stenosis, Crohn's disease) or gastrointestinal surgery(except for simple appendicitis surgery or hernia surgery or tooth extraction surgery) that may affect the absorption
3. Clinical laboratory test results showing the following values

   * ALT or AST > 2 times upper limit of normal range
4. Subject who has a history of regular alcohol consumption exceeding 210g/week within 6months of screening (1 glass of beer(5%)=10g, 1 glass of soju(20%)=8g, 1 glass of wine(12%)=12g)
5. Those taking other clinical trial drugs or bioequivalence test drugs within 3months before the first administration of clinical trial drug
6. Subject who has a systolic blood pressure of less than 100mmHg or more than 140mmHg or diastolic blood pressure of less than 60mmHg or more than 90mmHg of screening
7. Subject who has significant alcohol abuse or drug abuse within a year of screening
8. Those taking medication known to significantly induce or inhibit drug metabolizing enzymes within 30days prior to the first administration of clinical trial medication
9. More than 20 smokers per day within six months of screening
10. Those taking prescription or non-prescription drugs within 10days before the first administration of clinical trial medication
11. Those who donated whole blood within 2 months or those who donated the components within 1 month before the first administration of the clinical trial drug
12. Subject who has risk of serious or chronic medical, mental, or laboratory examinations that may increase the risk due to the administration of medicines for clinical trials and may interfere with the interpretation of test results
13. Patients who are known to be hypersensitive to the drug or its components
14. Patients with severe heart failure or heart failure(New York Heart Association(NYHA) Class 3, 4 heart patients)
15. Patients with hepatic impairment
16. Patients with a glomerular filtration rate(eGFR) less than 60ml/min/1.73m2, patients with end stage renal disease or dialysis
17. Patients with diabetic ketoacidosis, diabetic coma and total coma, patients with type 1 diabetes
18. Before and after surgery, severe infectious patients, severe trauma patients
19. Subjects with genetic problems such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
20. Pregnant and lactating women
21. Subject who is judged by the investigator to be ineligible to participate in the clinical trial

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2018-09-17 (Actual); Study Completion 2018-11-13 (Actual)

PRIMARY OUTCOMES:
(Part 1) AUCss,tau of D308 | Day 1, 3, 4 predose(0 hour) and Day 5 predose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours
  Area under the curve of D308 at steady state
(Part 1) Css,max of D308 | Day 1, 3, 4 predose(0 hour) and Day 5 predose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours
  Max Concentration of D308 at steady state
(Part 2) AUCss,tau of CKD-501 | Day 1, 3, 4 predose(0 hour) and Day 5 predose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours
  Area under the curve of CKD-501 at steady state
(Part 2) Css,max of CKD-501 | Day 1, 3, 4 predose(0 hour) and Day 5 predose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours
  Max Concentration of CKD-501 at steady state

SECONDARY OUTCOMES:
(Part 1) Css,min of D308 | Day 1, 3, 4 predose(0 hour) and Day 5 predose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours
  Min concentration of D308 at steady state
(Part 1) Css,av of D308 | Day 1, 3, 4 predose(0 hour) and Day 5 predose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours
  average concentration of D308 at steady state
(Part 1) Tss,max of D308 | Day 1, 3, 4 predose(0 hour) and Day 5 predose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours
  time of Max concentration of D308 at steady state
(Part 1) t1/2 of D308 | Day 1, 3, 4 predose(0 hour) and Day 5 predose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours
  half-life time of D308
(Part 1) CLss/F of D308 | Day 1, 3, 4 predose(0 hour) and Day 5 predose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours
  Apparent clearance of D308 at steady state
(Part 1) Vdss/F of D308 | Day 1, 3, 4 predose(0 hour) and Day 5 predose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours
  Apparent volume of distribution of D308 at steady state
(Part 1) Fluctuation[(Css,max-Css,min)/Css,av] of D308 | Day 1, 3, 4 predose(0 hour) and Day 5 predose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours
  Fluctuation concentration of D308 at steady state
(Part 1) Swing[(Css,max-Css,min)/Css,min] of D308 | Day 1, 3, 4 predose(0 hour) and Day 5 predose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours
  Swing concentration of D308 at steady state
(Part 2) Css,min of CKD-501 | Day 1, 3, 4 predose(0 hour) and Day 5 predose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours
  Min concentration of CKD-501 at steady state
(Part 2) Css,av of CKD-501 | Day 1, 3, 4 predose(0 hour) and Day 5 predose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours
  average concentration of CKD-501 at steady state
(Part 2) Tss,max of CKD-501 | Day 1, 3, 4 predose(0 hour) and Day 5 predose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours
  time of Max concentration of CKD-501 at steady state
(Part 2) t1/2 of CKD-501 | Day 1, 3, 4 predose(0 hour) and Day 5 predose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours
  half-life time of CKD-501
(Part 2) CLss/F of CKD-501 | Day 1, 3, 4 predose(0 hour) and Day 5 predose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours
  Apparent clearance of CKD-501 at steady state
(Part 2) Vdss/F of CKD-501 | Day 1, 3, 4 predose(0 hour) and Day 5 predose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours
  Apparent volume of distribution of CKD-501 at steady state
(Part 2) Fluctuation[(Css,max-Css,min)/Css,av] of CKD-501 | Day 1, 3, 4 predose(0 hour) and Day 5 predose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours
  Fluctuation concentration of CKD-501 at steady state
(Part 2) Swing[(Css,max-Css,min)/Css,min] of CKD-501 | Day 1, 3, 4 predose(0 hour) and Day 5 predose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours
  Swing concentration of CKD-501 at steady state

CONTACTS AND LOCATIONS:
Locations (1):
- Chonbuk National University Hospital, Jeonju, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jang K, Jeon JY, Moon SJ, Kim MG. Evaluation of the Pharmacokinetic Interaction Between Lobeglitazone and Dapagliflozin at Steady State. Clin Ther. 2020 Feb;42(2):295-304. doi: 10.1016/j.clinthera.2020.01.003. Epub 2020 Jan 25. PMID 31992459